CLINICAL TRIAL: NCT01394224
Title: A Single Site, Open-label, Randomized, Single-dose, Two-way Cross-over Study in Healthy Japanese Subjects to Evaluate the Bioequivalence, Safety & Tolerability of Levetiracetam Administered as an Oral Tablet or Intravenous Infusion
Brief Title: Bioequivalence Study of Levetiracetam Tablet and Intravenous Infusion in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: N01377; 2011-000827-34 (EudraCT Number)
Record Dates: First submitted 2011-07-12; First posted 2011-07-14 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers; Japanese
MeSH Terms: interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levetiracetam IV Infusion (1500 mg) (Experimental)
  Interventions: Drug: Levetiracetam
- Levetiracetam tablets (1500 mg) (Experimental)
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — Strength: 100 mg/mL Form: Concentrate for solution for infusion Frequency: Single dose
  Other Names: E-Keppra
  Arms: Levetiracetam IV Infusion (1500 mg)
Drug: Levetiracetam — Levetiracetam tablets Strength: 500 mg Form: Tablet Frequency: Single dose
  Other Names: E-Keppra
  Arms: Levetiracetam tablets (1500 mg)

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics(PK) and evaluate the bioequivalence of levetiracetam (LEV) following a single 15-minutes IV infusion of 1500 mg and a single oral dose(tablets) of 1500 mg in healthy Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese male and female volunteers with the age between 20 and 55 years old

Exclusion Criteria:

* Subject has participated or is participating in any other clinical studies of investigational drug or another IMP within the last 3 months
* Subject is not healthy (eg, taking any drug treatments, excessive amount of alcohol, cigarettes or caffeine, having any medical or emotional/psychological problems, a drug/alcohol abuse, having abnormal safety parameters)
* Subject is pregnant or lactating female.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Maximum drug concentration (Cmax) | Multiple sampling from 0 to 36 hours following single dose
Area under the plasma drug concentration versus time curve from hour 0 to the time with a last quantifiable level (AUCo-t) | Multiple sampling from 0 to 36 hours (could be less than 36 hours if the last quantifiable concentration is below limit of quantification), following single dose

SECONDARY OUTCOMES:
Time to reach maximum plasma concentration (tmax) | Multiple sampling from 0 to 36 hours following single dose
Plasma concentration at the end of infusion (C15' ) | At 15 minutes after termination of the15-minutes infusion
Area under the curve from 0 to infinity (AUC) | Multiple sampling from 0 to 36 hours following single dose
Mean resident time (MRT) | Multiple sampling from 0 to 36 hours following single dose
Terminal elimination half-life(t1/2) | Multiple sampling from 0 to 36 hours following single dose
First order terminal elimination rate constant (λz ) | Multiple sampling from 0 to 36 hours following single dose
Total body clearance after oral administration (CL/F) or after IV infusion (CL) | Multiple sampling from 0 to 36 hours following single dose
Volume of distribution after oral administration(Vz/F) or after IV infusion(Vz) | Multiple sampling from 0 to 36 hours following single dose

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- London, United Kingdom